CLINICAL TRIAL: NCT03641950
Title: Multi-center, Single Arm, Open-label, Phase IV Clinical Trial to Evaluate the Efficacy and Safety of Botulax® in Patients With Essential Blepharospasm
Brief Title: The Objective of This Study is to Evaluate the Efficacy and Safety of Botulax® in Patients With Essential Blepharospasm.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hugel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HG-BOT-IV3
Record Dates: First submitted 2018-08-19; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2016-03

CONDITIONS: Essential Blepharospasm
Keywords: Essential Blepharospasm
MeSH Terms: conditions — Benign essential blepharospasm | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Botulinum Toxin Type A (Botulax) (Experimental): Botulinum Toxin Type A (Botulax)
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Recommended initial dose to be intra-muscularly injected to the medial and contralateral pretarsal orbicularis oculi of the upper eyelid and the contralateral pretarsal orbicularis oculi of the lower eyelid is 1.25-2.5U (0.05ml ~ 0.1ml per site).
  Other Names: Botulax

SUMMARY:
The purpose of this study is evaluate the efficacy and safety of Botulax® in the treatment of Essential blepharospasm.

DETAILED DESCRIPTION:
Multi-center, single arm, open-label, Phase IV clinical trial to evaluate the efficacy and safety of Botulax® in Subjects with essential blepharospasm

ELIGIBILITY:
Inclusion Criteria:

1. Men and women at the age of 18 or older
2. Subjects diagnosed with essential blepharospasm with Jankovic Rating Scale (JRS) frequency and severity sum score ≥2 at screening
3. Individuals who agree to participate in the clinical study and voluntarily sign the written informed consent form
4. Subjects who are cooperative, have a good understanding of the clinical study, and can comply with study procedures until the end of the study

Exclusion Criteria:

1. Subjects who had received surgery such as orbicularis oculi resection or facial nerve block for the treatment of the study indication
2. Subjects with a history of hypersensitivity reactions to any of the components of the investigational product (botulinum toxins, serum albumin, etc.)
3. Subjects with secondary blepharospasm
4. Subjects with the hemifacial spasm
5. Subjects on treatment with muscle relaxants, benzodiazepines, anticholinergics, or benzamides who had changes in medication within 4 weeks prior to screening or have been on stable medication but are expected to have changes in medication while participating in the study
6. Subjects who administered any of the following drugs within 7 days prior to screening: drugs with muscle relaxation activity such as aminoglycoside antibiotics or other antibiotics (spectinomycin HCl, polypeptide antibiotics, tetracycline antibiotics, lincomycin antibiotics)
7. Subjects who administered medications similar to the investigational product (botulinum toxin type A) within 12 weeks
8. Subjects with systemic neuromuscular junction disorders: myasthenia gravis, Lambert-Eaton syndrome, or amyotrophic lateral sclerosis
9. Pregnant and lactating women
10. Women of childbearing potential who are planning to become pregnant within the next 3 months or are not using an appropriate method of contraception (contraceptive methods with an annual failure rate of less than 1% if used properly and continuously, including implant, injection, oral contraceptive, at least one barrier method such as intrauterine device [IUD], hormone IUD, abstinence, or vasectomized partner)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-01-07 (Actual)

PRIMARY OUTCOMES:
Total score change from baseline at 4 weeks post-injection of Jankovic Rating scale | At 4 weeks post-injection
  To evaluate the change of JRS (Jankovic Rating scale) score at 4 weeks post treatment based on baseline(0 week).
  JRS total score will be calculated as the sum (0~8) of two sub-scores of severity and frequency (0~4 each for severity and frequency) of blepharospasm.

SECONDARY OUTCOMES:
Total score change from baseline at 16 weeks post-injection of Jankovic Rating scale | At 0 weeks and 16 weeks post-injection
  To evaluate the change of JRS (Jankovic Rating scale) score at 16 weeks post treatment based on baseline(0 week)
Change from baseline at 4 weeks and 16 weeks of Disability Index | At 4 weeks and 16 weeks post-injection
  To evaluate the change of Blepharospasm Disability Index at 4 weeks and 16 weeks post treatment.
  Functional disability assessment scale will be assessed as functional disability score. Functional disability assessment scale consists of 6 daily activities (reading, watching television, household activities (cleaning, etc.), mobility, driving, work).
Global Response evaluated by investigator at 4 weeks and 16 weeks after post-injection | At 4 weeks and 16 weeks post-injection
  To evaluate the Investigator's assessment of global response at Weeks 4 and 16 after treatment.
  At Weeks 4 and 16 Visits after treatment, the investigator will assess global response on a 9-point scale from -4 (marked worsening) to +4 (Complete abolition of all signs and symptoms).
Change from baseline at 4 weeks and 16 weeks of WHO-Quality of Life(QOL) | At 4 weeks and 16 weeks post-injection
  To evaluate the change in WHO-Quality of Life (QoL) at Weeks 4 and 16 after treatment from baseline WHOQOL will be assessed by the brief Korean version of WHOQOL (WHOQOL-BREF). The Korean WHOQOL-BREF consists of a total of 26 subscales in 4 domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environment (8 items). Items in each subscale are in a range from 1 (not at all or very dissatisfied) to 5 (very much or very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Hugel, Seoul, Korea, South Korea